CLINICAL TRIAL: NCT04762134
Title: A Randomized Trial of Doxycycline Chemoprophylaxis for the Prevention of Sexually Transmitted Infections in Gay, Bisexual and Other Men Who Have Sex With Men (gbMSM)
Brief Title: Doxycycline Intervention for Bacterial STI ChemoprOphylaxis (DISCO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Troy Grennan (Other Government)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Jonathan Troy Grennan, Principal Investigator, British Columbia Centre for Disease Control
Organization: British Columbia Centre for Disease Control (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BritishCCDC3
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Bacterial Sexually Transmitted Diseases
Keywords: Sexually transmitted infections (STIs); Doxycycline; Pre-exposure prophylaxis (PrEP); Post-exposure prophylaxis (PEP); Gay, bisexual, men who have sex with other men (gbMSM)
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial; Sexually Transmitted Diseases; Homosexuality; Bisexuality | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomization with a 1:1 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STI PrEP arm (Experimental): doxycycline capsules 100mg orally daily for 12 months. Though the usual treatment dose of doxycycline is 100mg twice daily
  Interventions: Drug: Doxycycline Hyclate
- STI PEP arm (Experimental): doxycycline 200mg orally once within 24-72 hours following each sexual encounter deemed at risk (i.e. condomless anal or oral sex), to a maximum of six pills (i.e. 600 mg total) per week
  Interventions: Drug: Doxycycline Hyclate

INTERVENTIONS:
Drug: Doxycycline Hyclate — STI PrEP arm: doxycycline capsules 100mg orally daily for 12 months STI PEP arm: doxycycline 200mg orally once within 24-72 hours following each sexual encounter deemed at risk (i.e. condomless anal or oral sex), to a maximum of six pills (i.e. 600 mg total) per week

SUMMARY:
There is a growing epidemic of the bacterial sexually transmitted infections (STIs) syphilis, chlamydia and gonorrhea worldwide; similarly concerning trends have been noted in Canada, where increases of over 160% have been seen in bacterial STIs over the last decade. In Canada, gay, bisexual, and other men who have sex with men (gbMSM) - including those living with HIV - are disproportionately impacted by bacterial STIs5,6These dramatic increases in bacterial STIs, the potential development of serious complications including AMR, and waning effectiveness of the promotion of conventional STI prevention tools (e.g. condoms), signals the need for novel STI prevention strategies and tools to mitigate STI-related complications. A rigorous randomized controlled trial will be conducted to compare STI PrEP vs. STI PEP and definitively assess the efficacy, safety, antimicrobial resistance profiles and costs associated with doxycycline-based STI prevention.

DETAILED DESCRIPTION:
With the rising rates of STIs among gbMSM populations in Canada, there is an urgent need for novel interventions to prevent significant sequelae (e.g. neurosyphilis) and onward transmission of untreated infections. Despite longstanding public health efforts to encourage conventional strategies of STI prevention, gbMSM continue to bear the burden of syphilis which poses synergistic effects in the transmission of HIV. This study will add to this field through providing the first methodologically rigorous, prospective multicentre, open-label randomized controlled trial (RCT) of doxycycline-based STI PrEP (daily 100mg doxycycline) versus STI PEP (200mg doxycycline after exposure event) for the prevention of bacterial STIs among gbMSM over 15 months (60 weeks) of follow-up with adequate power to address drug efficacy in the prevention of bacterial STIs. Beyond the determination of efficacy, our trial will provide insight to the unique challenges of medication adherence through assessing the acceptability, tolerability and safety of therapy with doxycycline. This study aims to provide health care providers one additional tool to address the burden of STIs in populations with an increased likelihood of infection.

ELIGIBILITY:
Inclusion Criteria:

1. Males, ≥ 18 years of age;
2. Any sexual activity (i.e. oral sex, insertive or receptive anal sex, with or without a condom) with more than one male partner in the preceding 12 months;
3. Intention to remain sexually active with more than one male partner in the next 12 months;
4. At least one prior episode of a previously diagnosed and adequately treated syphilis, gonorrhea or chlamydia infection within 12 months prior to screening.

Exclusion Criteria:

1. Known allergy to doxycycline or tetracyclines;
2. Existing chronic or intermittent tetracycline or doxycycline use (e.g. for chronic osteomyelitis, acne).
3. Use of medications which could lower doxycycline levels, including barbiturates, phenytoin and carbamazepine.
4. Individuals currently using isotretinoin;
5. Any individual capable of becoming pregnant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gay, bisexual, and other men who have sex with men
Enrollment: 560 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma doxycycyline levels to determine efficacy of doxycycline chemoprophylaxis | 60 weeks
  To determine the efficacy of doxycycline chemoprophylaxis in preventing incident bacterial STI cases (syphilis, gonorrhea, and/or chlamydia, including LGV)

SECONDARY OUTCOMES:
Frequency of STIs over time | 60 weeks
  To describe frequency of syphilis, gonorrhea, and chlamydia incident infections among participants over the study period
Proportion of individuals reporting grade 3 or 4 adverse events in each study arm as assessed by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events | 60 weeks
  To determine the tolerability and safety of doxycycline chemoprophylaxis
Proportion of participants who report acceptability, community norms and partner attitudes of STI PrEP and PEP based on responses from questionnaires | 60 weeks
  To determine the acceptability of doxycycline chemoprophylaxis
Change in self-reported sexual activity defined as increases in condomless sexual acts and number of sexual partners based on responses from questionnaires | 60 weeks
  To evaluate the change in sexual behaviour reported by participants over the study period
Proportion of individuals with evidence of tetracycline class resistance in common flora (Staphylococcus aureus, Streptococcus pyogenes and Streptococcus pneumoniae) at 24 and 48 weeks. | Over 48 weeks
  To evaluate antimicrobial resistance in bacterial STIs and common commensal pathogens over study period
Proportion of cases with resistance to penicillins, tetracyclines or macrolides in syphilis, and tetracycline resistance in gonorrhea and chlamydia isolates taken from the anus, oral cavity or urethra. | Over 48 weeks
  To evaluate antimicrobial resistance in bacterial STIs and common commensal pathogens over study period
Proportion of individuals with adverse event-related study drug discontinuation in each study arm | Over 60 weeks
  To determine the tolerability and safety of doxycycline chemoprophylaxis
Rate of adherence to study treatment (STI PrEP vs. PEP) by participants. | Over 48 weeks
  To assess for superiority of doxycycline PrEP over PEP (if non-inferiority is shown)

CONTACTS AND LOCATIONS:
Overall Officials: Troy Grennan, MD, Principal Investigator — University of British Columbia
Locations (6):
- Canada (6):
  - Sheldon Chumir Centre, Calgary, Alberta
  - BC Centre for Disease Control, Vancouver, British Columbia
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
Our results will be targeted to four main groups of stakeholders: clinicians, public health, researchers, and community.The Community-Based Research Centre for Gay Men's Health, the Canadian AIDS Treatment Information Exchange (CATIE), and the AIDS Committee of Toronto will help facilitate KTE locally and nationally. We will disseminate our findings to a large, international audience of clinicians and public-health professionals by publishing in high-impact peer-reviewed journals.